CLINICAL TRIAL: NCT06812286
Title: TrackFrailty: Track to Prevent, Mitigate, and Reverse Frailty
Brief Title: TrackFrailty Project
Acronym: TrackFrailty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other); Health Sciences Research Centre (CICS-UBI) (Unknown); Reference Center for Active and Healthy Aging of the Interior Center Region (AgeINfuture) (Unknown); Universidad Pública de Navarra (Other); NavarraBiomed Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Mário Cardoso Marques, Full Professor, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCF/PR/SR24/57010031; LCF/PR/SR24/57010031 (Other Grant/Funding Number: "la Caixa" Foundation); UIDB/04045/2020 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology (FCT))
Record Dates: First submitted 2025-01-10; First posted 2025-02-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Frailty Syndrome
Keywords: Muscle Strength; Functional Performance; Cognitive Impairment; Depression; Anxiety; Social Support; Quality of Life; Resistance Training; Exercise; Nursing Homes; Aging
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: A statistician blinded to group allocation and the identity of the participants will analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Less-volume (Experimental): Three 10-week strength training cycles.
  Interventions: Other: Less-volume
- More-volume (Experimental): Three 10-week strength training cycles.
  Interventions: Other: More-volume
- Control (Other): Stretching exercises.
  Interventions: Other: Control

INTERVENTIONS:
Other: Less-volume — In the first 10-week cycle, the less-volume group will perform around 1500 repetitions per intervention. Participants will perform 1-3 sets of 4-7 repetitions per exercise with intensities ranging from 5% to 10% of body weight and 1-10 kg. Strength exercises will include chair squats, seated medicine ball throws, seated knee extensions, seated shoulder presses, standing calf raises, standing biceps curls, seated lateral raises, and chair stand + 4-meter walk. In the second and third 10-week training cycles, volume will increase by 20% with respect to the previous cycles. Two exercise physiologists will supervise training sessions.
  Arms: Less-volume
Other: More-volume — In the first 10-week cycle, the more-volume group will perform around 2000 repetitions per intervention. Participants will perform 1-3 sets of 6-10 repetitions per exercise with intensities ranging from 5% to 10% of body weight and 1-10 kg. Strength exercises will include chair squats, seated medicine ball throws, seated knee extensions, seated shoulder presses, standing calf raises, standing biceps curls, seated lateral raises, and chair stand + 4-meter walk. In the second and third 10-week training cycles, volume will increase by 20% with respect to the previous cycles. Two exercise physiologists will supervise training sessions.
  Arms: More-volume
Other: Control — Participants in the control group will undergo sham training twice weekly for 30 weeks, consisting of stretching exercises supervised by two exercise physiologists.
  Arms: Control

SUMMARY:
The TRACKFRAILTY project aims to answer the following main research questions:

i) What is the prevalence of physical frailty in individuals living in residential care facilities (RCF) from Portugal's Cova da Beira subregion (Interior Center Region)? ii) What factors best predict frailty status? iii) Is strength training effective in reversing physical frailty in RCF residents? iv) In the long term, what dose of strength training volume is needed to promote the most significant health benefits in frail RCF residents? Based on these research questions, the TRACKFRAILTY project aims to quantify the prevalence of frailty in Portuguese RCF residents from the Cova da Beira subregion and analyze the effects of long-term strength training with different volumes on reversing physical frailty.

DETAILED DESCRIPTION:
The TRACKFRAILTY project will consist of two primary research activities. Activity one will be a cross-sectional study to quantify the prevalence of physical frailty in residential care facility (RCF) residents from Portugal's Cova da Beira subregion (Interior Center Region). Activity two will be a randomized controlled trial to compare different strength training volumes for reversing frailty in RCF residents.

The prevalence study will include a representative sample of RCF residents from Portugal's Cova da Beira subregion. The investigators will use a comprehensive recruitment strategy, including contacts and meetings with the technical directors of several RCFs from the Cova da Beira subregion. Participants must comply with the inclusion criteria to make part of the study, namely men or women aged 50 and above residing in RCFs in Cova da Beira, capable of collaborating with the research team members, and giving written or oral informed consent. Exclusion criteria will comprise individuals with severe dementia (inability to speak or communicate with permanent care and assistance) and hospitalized and bedridden individuals.

After recruitment, the investigators will implement an evaluation protocol in two parts. The first part will include the collection of i) sociodemographic data, ii) diseases, iii) medications, iv) smoking status and alcohol consumption, v) self-perceived health-related quality of life, vi) self-reported unintentional weight loss, vii) falls history (last 12 months); viii) disability level, ix) self-reported exhaustion, x) physical activity level, xi) cognitive function, xii) emotional state, and xiii) relational/social aspects. The second part will include the collection of i) hemodynamic data, ii) anthropometric data, iii) lower extremity function data, and iv) upper extremity function data. The investigators will assess frailty using Fried's criteria (self-reported unintentional weight, self-reported exhaustion, low physical activity, muscle weakness, and slowness). Individuals with 3-5 criteria will be considered frail, 1-2 pre-frail, and 0 non-frail. Frail and pre-frail individuals will be invited to participate in the randomized controlled trial.

Research activity two will be a randomized, single-blind, three-arm (two experimental groups and one control group), parallel-group study of 30 weeks. The investigators will randomly assign the participants into three groups: less-volume (LV), more-volume (MV), and control (CG). The CG will perform stretching exercises supervised by two exercise physiologists during the intervention (two sessions per week). The LV and MV groups will undergo three 10-week strength training cycles, each with two weekly sessions. In the first cycle, LV will perform around 1500 total repetitions, while MV will perform around 2000. In the second and third cycles, the volume will increase by 20% with reference to the previous cycles in both experimental groups. Training frequency, exercises, and intensities will be the same in both groups. In brief, participants will perform 1-3 sets per exercise of 4-7 repetitions (LV) or 6-10 repetitions (MV) with intensities ranging from 5% to 10% of body weight and 1-10 kg. Strength exercises will include chair squats, seated medicine ball throws, seated knee extensions, seated shoulder presses, standing calf raises, standing biceps curls, seated lateral raises, and chair stand + 4-meter walk.

The investigators will administer the evaluation protocol described in research activity one before the first 10-week training cycle and after the first, second, and third 10-week training cycles. The primary outcome measure will be the frailty phenotype (Fried's criteria). The secondary outcome measures will include physical tests, cognitive function, emotional state, relational aspects, health-related quality of life, falls, feasibility, and safety. A statistician will analyze the data following an intention-to-treat and per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women residing in residential care facilities (RFC) from the Cova da Beira subregion of Portugal
* Non-frail, pre-frail, and frail individuals (prevalence study)
* Pre-frail and frail individuals (randomized controlled trial)
* Capable of collaborating with the research team members
* Capable of giving written or oral informed consent

Exclusion Criteria:

* Severe dementia (inability to speak or communicate with permanent care and assistance)
* Hospitalized and bedridden individuals

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Frailty phenotype | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  Fried's criteria will be used to assess frailty (unintentional weight loss, exhaustion, low physical activity, slowness, and muscle weakness).

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The SPPB consists of three tests (balance, 4-meter walking, and 5-repetition sit-to-stand), and the score ranges from 0-12, with lower scores indicating worse physical function.
10-meter walking test | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  Participants will walk 10 m in a linear path, and time (s) will be measured.
6-minute walking test | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  Participants will walk back and forth on 10 to 15 m paths for 6 minutes, and the total distance (m) covered during the stipulated time will be measured.
Handgrip strength | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  A handheld dynamometer will be used to measure handgrip strength (seated position).
1-kg medicine ball throw | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  In a seated position, participants will throw the 1-kg medicine ball, and the distance (m) will be measured using a tape measure.
Montreal Cognitive Assessment (MoCA) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The Montreal Cognitive Assessment (MoCA) will be used to detect cognitive impairment. It assesses different cognitive domains, such as memory, executive functioning, attention, language, visuospatial, and orientation, and the maximum score is 30 (lower scores indicate different cognitive impairment levels).
Satisfaction With Life Scale (SWLS) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The Satisfaction with Life Scale (SWLS) consists of five items, each scored on a 7-point Likert scale ranging from "strongly disagree" to "strongly agree". The SWLS score is the sum of the item scores, ranging from 5 (lowest satisfaction) to 35 (highest satisfaction).
Geriatric Depression Scale (GDS) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The Geriatric Depression Scale (GDS) consists of 30 questions answered with "yes" or "no". The GDS score is the sum of all answers, with higher scores indicating higher depression levels.
Geriatric Anxiety Inventory (GAI) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The Geriatric Anxiety Inventory (GAI) consists of 20 questions answered with "yes" or "no". The GAI score is the sum of all answers, with higher scores indicating the presence of anxiety.
Brief 2-Way Social Support Scale (SSS) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The Brief 2-Way Social Support Scale (SSS) consists of 12 items to measure four dimensions of social support (giving emotional support, receiving emotional support, giving instrumental support, and receiving instrumental support). Each item is scored on a 6-point Likert scale ranging from "never" to "always".
6-item De Jong Gierveld Loneliness Scale (DJGLS-6) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The 6-item De Jong Gierveld Loneliness Scale (DJGLS-6) has three statements about emotional loneliness (items 1, 2, and 3) and three statements about social loneliness (items 4, 5, and 6). Each item is scored with "yes", "more or less", and "no". In items 1, 2, and 3, "yes" and "more or less" are classified with 1 and "no" with 0. In items 4, 5, and 6, yes" is classified with 0, and "more or less" and "no" are classified with 1. The DJGLS-6 score ranges from 0 to 6, with lower scores indicating "least lonely".
Health-Related Quality of Life 36-Item Short Form Survey (SF-36) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The SF-36 consists of 36 items to assess physical (4 scales: physical functioning, role-physical, bodily pain, and general health) and mental health (4 scales: vitality, social functioning, role-emotional, and emotional well-being). First, each item is scored with a Likert scale or "yes" or "no" answers. Afterward, each item is rated on a scale of 0 to 100. The higher the scores in each scale, the higher the perception of health-related quality of life.
Falls | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The number of falls during the intervention will be registered.
Recruitment, Retention, and Adherence Rates (Feasibility) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The recruitment, retention, and adherence rates will be calculated to analyze the feasibility of the intervention.
Incidence of Adverse Events during Intervention (Safety) | Baseline and after 10, 20, and 30 weeks of intervention (4 time points).
  The number of adverse events (an undesirable outcome during the intervention that may or may not be related to it) will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Mário C Marques, PhD, Principal Investigator — University of Beira Interior
Locations (6):
- Portugal (6):
  - Santa Casa da Misericórdia da Covilhã, Covilha, Castelo Branco District
  - Centro Social Nossa Senhora da Conceição, Covilha, Castelo Branco District
  - Lar de São José, Covilha, Castelo Branco District
  - Associação Centro Social Sagrado Coração Maria, Covilha, Castelo Branco District
  - Santa Casa da Misericórdia do Fundão, Fundão, Castelo Branco District
  - Centro Social Vales do Rio, Covilha, Cas

IPD SHARING:
Plan to Share IPD: No